CLINICAL TRIAL: NCT04159909
Title: Using Transcutaneous Auricular Vagus Nerve Stimulation to Treat Acute Alcohol Withdrawal
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study site, detoxification unit at South Oaks Hospital, was closed/partially open. Northwell addiction has been unable to provide any projected/workable plan(s).
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-0576
Record Dates: First submitted 2019-11-05; First posted 2019-11-12 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Alcohol Withdrawal; Alcohol Use Disorder
Keywords: vagus nerve stimulation (VNS), non-invasive intervention
MeSH Terms: conditions — Alcoholism | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized, single-blinded Treatment vs sham
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- VNS transcutaneous stimulation (Experimental): 5 minutes of stimulation (VNS) twice a day for 4 days. Patients will receive transcutaneous stimulation (30 Hz, 300 msec.) on the auricular branch of the vagus nerve 5 minutes twice a day for 4 days. Due to the theoretical risk that right vagus nerve stimulation could affect the heart, and to ensure consistency of the intervention, all subjects randomized to receive transcutaneous vagus nerve stimulation will receive stimulation of the auricular branch of the left vagus nerve. The subject will be blinded to their treatment arm.
  The device to be used will include a handheld electrical pulse generator and a pair of electrodes to be placed at the ear for stimulation. The specific target at the ear will be the auricular branch of the vagus nerve, which innervates the skin of a specific ear area termed "Cymba Concha". Electrodes will be placed on this area to provide stimulation to the auricular branch of the afferent vagus nerve.
  Interventions: Device: Transcutaneous Nerve Stimulation
- Sham stimulation (Sham Comparator): 5 minutes of sham stimulation (no electrical stimulation) twice a day for 4 days Patients will receive sham stimulation on the auricular branch of the vagus nerve 5 minutes twice a day for 4 days.
  The subject will be blinded to their treatment arm. The specific target at the ear will be the auricular branch of the vagus nerve, which innervates the skin of a specific ear area termed "Cymba Concha". Electrodes will be placed on this area to provide sham stimulation (no electrical current) to the auricular branch of the afferent vagus nerve.
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Transcutaneous Nerve Stimulation — 510(K) number: K110390 vagus nerve for 5 minutes twice a day for 4 consecutive days
  Arms: VNS transcutaneous stimulation
Device: Sham Stimulation — sham stimulation (no electrical current) for 5 minutes twice a day for 4 consecutive days
  Arms: Sham stimulation

SUMMARY:
The purpose of this study is to see if stimulation of the vagus nerve via a non-invasive device placed behind external ear can reduce physical and psychological discomfort during acute alcohol withdrawal in patients with alcohol use disorder when people just stop drinking alcohol and in detoxification stage.

DETAILED DESCRIPTION:
The management of acute alcohol withdrawal is a clinical challenge, in part because there are limited medications available for the condition and the majority of the medications are controlled substances, which may cause significant adverse effects and can be potentially addictive.

The rationale for using transcutaneous auricular VNS (taVNS) on a specific target area of the ear is based on anatomical studies suggesting that this area is the only place on the human body surface where there is afferent vagus nerve distribution (Mercante et al., 2018). Therefore, direct stimulation of the afferent nerve fibers on the ear can produce an effect similar to that by implanted device-generated VNS yet without the need of surgical intervention. Although taVNS has not been tested for treatment of AUD, it interestingly appears to be very similar to auricular acupuncture that has been widely used for AUD. However, acupuncture needs to be administered by medical providers who have undergone long trainings and own special licensure, which is usually unavailable in acute detoxification units where patients receive treatment for acute alcohol withdrawal.

The pilot study will enroll 70 evaluable subjects who are in inpatient detoxification unit randomized to receive single-blind treatment with vagus nerve stimulation or sham stimulation (1:1, VNS: sham). Evaluable subjects are those who complete stimulations (VNS) or sham 5 minutes twice a day for 4 days.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-65 years (men and women);
2. primary current diagnosis of DSM-V Alcohol Use Disorder as indicated at admission;
3. being admitted to inpatient detoxification unit;
4. no evidence of significant cognitive impairment with a mini mental state examination (MMSE; Folstein et al., 1975) score > 22;
5. able and willing to give written informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

1. current DSM-V substance use disorders (other than tobacco / cannabis/ alcohol);
2. serious psychiatric illnesses, e.g. psychotic disorders or bipolar disorder
3. severe medical illnesses, present or history of, e.g. hepatic encephalopathy, delirium
4. history of significant medical problems associated with drinking including seizures;
5. pregnancy;
6. severe intellectual/cognitive deficits due to Korsakoff's syndrome, dementia, head injury, or others
7. treatment with an anti-cholinergic medication, including over the counter medications,
8. implantable electronic devices such as pacemakers, defibrillators, hearing aids, cochlear implants or deep brain stimulators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-31 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
The primary clinical outcome is the reduction of the alcohol withdrawal symptoms assessed by the Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar) | 3 months after completion of pilot study (enrollment)
  The primary clinical endpoint is the alcohol withdrawal symptoms assessed by the Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar) (Sullivan, Sykora, Schneiderman, Naranjo, & Sellers, 1989) as well as the amount and frequency of as needed comfort medications (benzodiazepines, e.g., Chlordiaxepoxide, Lorazepam) used from day 1 to day 4 by the participants in acute detoxification inpatient unit treated with VNS compared to subjects receiving sham stimulation.

OTHER OUTCOMES:
Assesssment of change of neruroinflammatory reflex by measurement of blood levels of cytokines following VNS treatment for acute alcohol withdrawal | 6 months after completion of pilot study (enrollment)
  The mechanistic endpoints accompanying this protocol will evaluate potential effects of VNS on inflammatory markers and cytokines known to be involved with AUD. 8 ml venous whole blood from participants will be collected on Day 1 before receiving any VNS or sham treatment and on Day 5 after completing all 8 treatments. Serum and plasma from 8cc of whole blood will be collected, stored in aliquots at -20∙C. Serum levels of potential inflammatory markers and markers regulated by the alpha-7nAChR will be determined, including levels of pro-inflammatory cytokines, TNF, HMGB1, IL-6, Il1B, IFNα and IL10 which are known to be elevated in patients with AUD.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C Chen, MD, PhD, Principal Investigator — Northwell Health
Locations (1):
- Feinstein Institutes for Medical Research, Northwell Health, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mercante B, Ginatempo F, Manca A, Melis F, Enrico P, Deriu F. Anatomo-Physiologic Basis for Auricular Stimulation. Med Acupunct. 2018 Jun 1;30(3):141-150. doi: 10.1089/acu.2017.1254. PMID 29937968
- [Background] Kreuzer PM, Landgrebe M, Husser O, Resch M, Schecklmann M, Geisreiter F, Poeppl TB, Prasser SJ, Hajak G, Langguth B. Transcutaneous vagus nerve stimulation: retrospective assessment of cardiac safety in a pilot study. Front Psychiatry. 2012 Aug 7;3:70. doi: 10.3389/fpsyt.2012.00070. eCollection 2012. PMID 22891061
- [Background] Baker TE, Chang G. The use of auricular acupuncture in opioid use disorder: A systematic literature review. Am J Addict. 2016 Dec;25(8):592-602. doi: 10.1111/ajad.12453. Epub 2016 Nov 2. PMID 28051842
- [Background] Sullivan JT, Sykora K, Schneiderman J, Naranjo CA, Sellers EM. Assessment of alcohol withdrawal: the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar). Br J Addict. 1989 Nov;84(11):1353-7. doi: 10.1111/j.1360-0443.1989.tb00737.x. PMID 2597811